CLINICAL TRIAL: NCT07258199
Title: Transarterial Chemoembolization With Bleomycin: A Promising Treatment of Giant Nodular Goiter
Brief Title: TACE Treats Nodular Goiter
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TACE treats nodular goiter
Record Dates: First submitted 2025-09-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Nodular Goiter
Keywords: Transarterial chemoembolization; Giant nodular goiter; Bleomycin; Drug-loaded microspheres
MeSH Terms: conditions — Goiter, Nodular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE (Experimental)
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — TACE, 15,000U bleomycin and 200-400μm drug-loaded microspheres

SUMMARY:
transarterial bleomycin chemoembolization represents a novel minimally invasive therapeutic approach for the management of giant nodular goiter.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria: thyroid enlargement, mostly painless, with compressive symptoms (such as dysphagia, dyspnea) being less common; thyroid function is mostly normal, and a small number may be accompanied by hyperthyroidism or hypothyroidism.
* Imaging examinations: ultrasound shows multiple solid or cystic-solid nodules with clear boundaries and no malignant signs such as microcalcification and a vertical-to-horizontal diameter ratio >1.
* Pathological criteria: follicular epithelial cell hyperplasia, no nuclear atypia, and no malignant cellular characteristics (such as mitotic figures, infiltrative growth, etc.). In this study, a thyroid goiter with at least one diameter exceeding 4 cm was considered a giant goiter

Exclusion Criteria:

* abnormal coagulation profiles;
* hepatic or renal impairment;
* allergy to contrast media;
* refusal of interventional therapy and requirement for surgical treatment or other therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
volume | 1-, 3-, 6-, 12-month follow up
  Lesion volume measurement on contrast-enhanced CT

SECONDARY OUTCOMES:
longest diameter | 1-, 3-, 6-, 12-month follow-up
  Measurement of the longest lesion diameter on contrast-enhanced CT
lesion shrinkage | 1-, 3-, 6-, 12-month follow-up

OTHER OUTCOMES:
postoperative complications | 1-, 3-, 6-, 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes